CLINICAL TRIAL: NCT00481546
Title: Phase I Trial of Ocular Subretinal Injection of a Recombinant Adeno-Associated Virus (rAAV2-CBSB-hRPE65) Gene Vector to Patients With Retinal Disease Due to RPE65 Mutations (Clinical Trials of Gene Therapy for Leber Congenital Amaurosis)
Brief Title: Phase I Trial of Gene Vector to Patients With Retinal Disease Due to RPE65 Mutations
Acronym: LCA
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 547233; Grant: 1 U10 EY017280-01;; UP IRB: 804582;; UP IBC: 06-105;; UF GCRC: 675;; UF IBC RD: 2795;; WIRB: 20061300
Record Dates: First submitted 2007-05-31; First posted 2007-06-01 (Estimated); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Amaurosis of Leber; Retinal Diseases
Keywords: Leber congenital amaurosis; LCA; RPE65; Retinal disease due to RPE65 mutations; RPE65-associated Leber congenital amaurosis
MeSH Terms: conditions — Retinal Diseases; Leber Congenital Amaurosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental (Experimental): All clinical trial subjects received the same vector.
  Interventions: Genetic: rAAV2-CBSB-hRPE65

INTERVENTIONS:
Genetic: rAAV2-CBSB-hRPE65 — One or two, uniocular, subretinal injections; relative doses: 0.3X (Cohort 1), 0.6X (Cohort 2), 0.45X (Cohort 3), 0.9X (Cohorts 4 and 5)

SUMMARY:
A recombinant adeno-associated virus serotype 2 (rAAV2) vector has been altered to carry the human RPE65 (hRPE65) gene. This vector has been shown to restore vision in animal models that resemble human RPE65-associated Leber congenital amaurosis (LCA), an incurable retinal degeneration that causes severe vision loss. The proposed study is an open label, Phase I clinical trial of subretinal rAAV2-CBSB-hRPE65 administration to individuals with RPE65-associated retinal disease. Five cohorts will be included in this trial. Cohorts 1, 2 and 4 will consist of individuals 18 years of age and older. Cohorts 3 and 5 will consist of individuals between the ages of 8 and 17, inclusive. Enrollment in Cohorts 3 and 5 will begin only after confirming the safety of rAAV2-CBSB-hRPE65 administration in the older groups of participants. This trial will lead to a greater understanding of the safety and thereby potential value of gene transfer in RPE65-associated retinal disease and will have implications for other forms of retinal degenerative disease amenable to this type of intervention.

The goal of this clinical trial is to determine the safety of uniocular subretinal administration of rAAV2-CBSB-hRPE65 in individuals with RPE65-associated retinal disease. Ocular and systemic toxicity will be assessed prior to and following vector administration to determine if there are adverse changes that may be associated with vector administration.

ELIGIBILITY:
Inclusion Criteria:

* RPE65-associated retinal disease (two disease-causing RPE65 mutations);
* Clinical diagnosis of Leber congenital amaurosis (LCA)/early-onset retinal degeneration (EORD) and of severely impaired visual and retinal function, and best corrected visual acuity of 20/40 or worse in the study eye;
* Ability to perform tests of visual and retinal function;
* Visible photoreceptor layer on a standard OCT scan;
* Good general health;
* Ability to comply with research procedures;
* Specific for Cohorts 1, 2 and 4: 18 years of age and older;
* Specific for Cohorts 3 and 5: Between 8 and 17 years of age, inclusive.

Exclusion Criteria:

* AAV antibody titers greater than two standard deviations above normal at baseline;
* Humoral immune deficiency as evidenced by low tetanus toxoid IgG antibody titers;
* Pre-existing eye conditions that would preclude the planned surgery or interfere with the interpretation of study endpoints or surgical complications;
* Complicating systemic diseases;
* Use of anti-platelet agents that may alter coagulation within 7 days prior to study agent administration;
* Use of immunosuppressive medications;
* Pregnancy or breastfeeding;
* Individuals (males and females) of childbearing potential who are unwilling to use effective contraception;
* Any condition that would prevent a subject from completing follow-up examinations during the course of the study;
* Any condition that makes the subject unsuitable for the study;
* Current, or recent participation, in any other research protocol involving investigational agents or therapies;
* Recent receipt of an investigational biologic therapeutic agent.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2007-07; Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The primary safety endpoint in this trial is the standard ocular examination. Toxicity will also be assessed by measurement of vision, hematology and serum chemistries, assays for vector genomes, reported subject history of symptoms and adverse events. | 15 years

SECONDARY OUTCOMES:
Visual function will be quantified prior to and after vector administration in order to determine whether vector administration affects visual function. | 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Samuel G. Jacobson, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Shands Children's Hospital, University of Florida, Gainesville, Florida
  - Scheie Eye Institute, University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Jacobson SG, Boye SL, Aleman TS, Conlon TJ, Zeiss CJ, Roman AJ, Cideciyan AV, Schwartz SB, Komaromy AM, Doobrajh M, Cheung AY, Sumaroka A, Pearce-Kelling SE, Aguirre GD, Kaushal S, Maguire AM, Flotte TR, Hauswirth WW. Safety in nonhuman primates of ocular AAV2-RPE65, a candidate treatment for blindness in Leber congenital amaurosis. Hum Gene Ther. 2006 Aug;17(8):845-58. doi: 10.1089/hum.2006.17.845. PMID 16942444
- [Background] Jacobson SG, Acland GM, Aguirre GD, Aleman TS, Schwartz SB, Cideciyan AV, Zeiss CJ, Komaromy AM, Kaushal S, Roman AJ, Windsor EA, Sumaroka A, Pearce-Kelling SE, Conlon TJ, Chiodo VA, Boye SL, Flotte TR, Maguire AM, Bennett J, Hauswirth WW. Safety of recombinant adeno-associated virus type 2-RPE65 vector delivered by ocular subretinal injection. Mol Ther. 2006 Jun;13(6):1074-84. doi: 10.1016/j.ymthe.2006.03.005. Epub 2006 Apr 27. PMID 16644289
- [Background] Acland GM, Aguirre GD, Bennett J, Aleman TS, Cideciyan AV, Bennicelli J, Dejneka NS, Pearce-Kelling SE, Maguire AM, Palczewski K, Hauswirth WW, Jacobson SG. Long-term restoration of rod and cone vision by single dose rAAV-mediated gene transfer to the retina in a canine model of childhood blindness. Mol Ther. 2005 Dec;12(6):1072-82. doi: 10.1016/j.ymthe.2005.08.008. Epub 2005 Oct 14. PMID 16226919
- [Background] Jacobson SG, Aleman TS, Cideciyan AV, Sumaroka A, Schwartz SB, Windsor EA, Traboulsi EI, Heon E, Pittler SJ, Milam AH, Maguire AM, Palczewski K, Stone EM, Bennett J. Identifying photoreceptors in blind eyes caused by RPE65 mutations: Prerequisite for human gene therapy success. Proc Natl Acad Sci U S A. 2005 Apr 26;102(17):6177-82. doi: 10.1073/pnas.0500646102. Epub 2005 Apr 18. PMID 15837919
- [Background] Acland GM, Aguirre GD, Ray J, Zhang Q, Aleman TS, Cideciyan AV, Pearce-Kelling SE, Anand V, Zeng Y, Maguire AM, Jacobson SG, Hauswirth WW, Bennett J. Gene therapy restores vision in a canine model of childhood blindness. Nat Genet. 2001 May;28(1):92-5. doi: 10.1038/ng0501-92. PMID 11326284
- [Background] Jacobson SG, Aleman TS, Cideciyan AV, Heon E, Golczak M, Beltran WA, Sumaroka A, Schwartz SB, Roman AJ, Windsor EA, Wilson JM, Aguirre GD, Stone EM, Palczewski K. Human cone photoreceptor dependence on RPE65 isomerase. Proc Natl Acad Sci U S A. 2007 Sep 18;104(38):15123-8. doi: 10.1073/pnas.0706367104. Epub 2007 Sep 11. PMID 17848510
- [Background] Jacobson SG, Aleman TS, Cideciyan AV, Roman AJ, Sumaroka A, Windsor EA, Schwartz SB, Heon E, Stone EM. Defining the residual vision in leber congenital amaurosis caused by RPE65 mutations. Invest Ophthalmol Vis Sci. 2009 May;50(5):2368-75. doi: 10.1167/iovs.08-2696. Epub 2008 Dec 30. PMID 19117922
- [Background] Jacobson SG, Cideciyan AV, Aleman TS, Sumaroka A, Windsor EA, Schwartz SB, Heon E, Stone EM. Photoreceptor layer topography in children with leber congenital amaurosis caused by RPE65 mutations. Invest Ophthalmol Vis Sci. 2008 Oct;49(10):4573-7. doi: 10.1167/iovs.08-2121. Epub 2008 Jun 6. PMID 18539930
- [Background] Jacobson SG, Cideciyan AV. Treatment possibilities for retinitis pigmentosa. N Engl J Med. 2010 Oct 21;363(17):1669-71. doi: 10.1056/NEJMcibr1007685. No abstract available. PMID 20961252
- [Background] Cideciyan AV. Leber congenital amaurosis due to RPE65 mutations and its treatment with gene therapy. Prog Retin Eye Res. 2010 Sep;29(5):398-427. doi: 10.1016/j.preteyeres.2010.04.002. Epub 2010 Apr 24. PMID 20399883
- [Result] Cideciyan AV, Aleman TS, Boye SL, Schwartz SB, Kaushal S, Roman AJ, Pang JJ, Sumaroka A, Windsor EA, Wilson JM, Flotte TR, Fishman GA, Heon E, Stone EM, Byrne BJ, Jacobson SG, Hauswirth WW. Human gene therapy for RPE65 isomerase deficiency activates the retinoid cycle of vision but with slow rod kinetics. Proc Natl Acad Sci U S A. 2008 Sep 30;105(39):15112-7. doi: 10.1073/pnas.0807027105. Epub 2008 Sep 22. PMID 18809924
- [Result] Hauswirth WW, Aleman TS, Kaushal S, Cideciyan AV, Schwartz SB, Wang L, Conlon TJ, Boye SL, Flotte TR, Byrne BJ, Jacobson SG. Treatment of leber congenital amaurosis due to RPE65 mutations by ocular subretinal injection of adeno-associated virus gene vector: short-term results of a phase I trial. Hum Gene Ther. 2008 Oct;19(10):979-90. doi: 10.1089/hum.2008.107. PMID 18774912
- [Result] Cideciyan AV, Hauswirth WW, Aleman TS, Kaushal S, Schwartz SB, Boye SL, Windsor EA, Conlon TJ, Sumaroka A, Pang JJ, Roman AJ, Byrne BJ, Jacobson SG. Human RPE65 gene therapy for Leber congenital amaurosis: persistence of early visual improvements and safety at 1 year. Hum Gene Ther. 2009 Sep;20(9):999-1004. doi: 10.1089/hum.2009.086. PMID 19583479
- [Result] Cideciyan AV, Hauswirth WW, Aleman TS, Kaushal S, Schwartz SB, Boye SL, Windsor EA, Conlon TJ, Sumaroka A, Roman AJ, Byrne BJ, Jacobson SG. Vision 1 year after gene therapy for Leber's congenital amaurosis. N Engl J Med. 2009 Aug 13;361(7):725-7. doi: 10.1056/NEJMc0903652. No abstract available. PMID 19675341
- [Result] Jacobson SG, Cideciyan AV, Ratnakaram R, Heon E, Schwartz SB, Roman AJ, Peden MC, Aleman TS, Boye SL, Sumaroka A, Conlon TJ, Calcedo R, Pang JJ, Erger KE, Olivares MB, Mullins CL, Swider M, Kaushal S, Feuer WJ, Iannaccone A, Fishman GA, Stone EM, Byrne BJ, Hauswirth WW. Gene therapy for leber congenital amaurosis caused by RPE65 mutations: safety and efficacy in 15 children and adults followed up to 3 years. Arch Ophthalmol. 2012 Jan;130(1):9-24. doi: 10.1001/archophthalmol.2011.298. Epub 2011 Sep 12. PMID 21911650
- [Derived] Jacobson SG, Cideciyan AV, Roman AJ, Sumaroka A, Schwartz SB, Heon E, Hauswirth WW. Improvement and decline in vision with gene therapy in childhood blindness. N Engl J Med. 2015 May 14;372(20):1920-6. doi: 10.1056/NEJMoa1412965. Epub 2015 May 3. PMID 25936984
- [Derived] Cideciyan AV, Aguirre GK, Jacobson SG, Butt OH, Schwartz SB, Swider M, Roman AJ, Sadigh S, Hauswirth WW. Pseudo-fovea formation after gene therapy for RPE65-LCA. Invest Ophthalmol Vis Sci. 2014 Dec 23;56(1):526-37. doi: 10.1167/iovs.14-15895. PMID 25537204